CLINICAL TRIAL: NCT06289543
Title: The Effect of A Newly Formulated Preoperative Oral Carbohydrate Solution on Gastric Emptying, Postoperative Nausea and Vomiting and Stress Response
Brief Title: Preoperative Oral Carbohydrate on Gastric Emptying
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Emine Şeyda Teloğlu, Physician, Department of Anesthesiology, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BVU-ESTELOGLU
Record Dates: First submitted 2024-01-29; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Vomit Aspiration; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Water

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Starvation (No Intervention): Fasting for 6-8 hours before the operation
- Water (Active Comparator): drink 400ml of water 2 hours before the operation
  Interventions: Dietary Supplement: Preoperative carbohydrate solution
- oral carbohydrate (Active Comparator): drink 400ml of solution 2 hours before the operation
  Interventions: Dietary Supplement: Preoperative carbohydrate solution

INTERVENTIONS:
Dietary Supplement: Preoperative carbohydrate solution — water and solution will be given to patients to drink 2 hours before the operation
  Other Names: Water
  Arms: Water; oral carbohydrate

SUMMARY:
The current preoperative fasting guidelines recommend, applying preoperative carbohydrate solution 2 hours before the operation to minimize prolonged fasting time potential negative effects and improve patient comfort. Fasting after midnight before the operation day is a widespread practice. The major obstacle to preoperative carbohydrate solutions becoming prevalent and extremely long fasting time is the limited product; which is proven safe and efficient, and unavailable in several countries. In this study, our objective is to analyze the gastric volume, preoperative anxiety, stress response, postoperative insulin resistance, and postoperative nausea and vomiting by utilizing a low osmolality oral carbohydrate solution prepared with ginger and melissa.

DETAILED DESCRIPTION:
The current preoperative fasting guidelines recommend, applying preoperative carbohydrate solution 2 hours before the operation to minimize prolonged fasting time potential negative effects and improve patient comfort. Fasting after midnight before the operation day is a widespread practice. The major obstacle to preoperative carbohydrate solutions becoming prevalent and extremely long fasting time is the limited product; which is proven safe and efficient, and unavailable in several countries. In this study, our objective is to analyze the gastric volume, preoperative anxiety, stress response, postoperative insulin resistance, and postoperative nausea and vomiting by utilizing a low osmolality oral carbohydrate solution prepared with ginger and melissa.

109 patients who underwent elective laparoscopic cholecystectomy, aged 18-65 years, and ASA physical state 1-2 were included in the study. The patients were divided into 3 groups: Group A, who would not eat anything 6-8 hours before the operation, Group S, who drank 400 ml of water 2 hours before the operation, and Group K, which drank 400 ml preoperative oral carbohydrate solution (PreOKH) 2 hours before the operation. Before induction of anesthesia (T1), patients' antral gastric cross-sectional area (GKA) and gastric volume (GV) were evaluated by gastric ultrasound. The preoperative anxiety level of the patients was determined by the State-Trait Anxiety Inventory (STAl) before the operation (T1), and the symptoms affecting the preoperative patient comfort parameters (thirst, hunger, dry mouth, fatigue) were measured 2 hours before the operation (T0) and before the induction (T1) evaluated with the visual analog scale (VAS). Postoperative nausea and vomiting (PONV) and postoperative pain levels were recorded. Blood glucose, insulin, and cortisol levels of the patients were measured 2 hours before the operation (T0), before induction (T1), and postoperative 2nd hour (T3)

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Elective laparoscopic cholecystectomy planned under general anesthesia
* American Society of Anesthesiologists (ASA) class I-II physical condition

Exclusion Criteria:

Patients with gastroesophageal reflux and gastrointestinal motility disorders diabetes mellitus Mental retardation, previous neurological disease symptoms (syncope, dementia, Alzheimer, etc.) Chronic alcoholism Difficult Intubation Patients with ASA physical status classes ≥III Patients with a body mass index of 35 and above History of Meniere and motion sickness Presence of previous history of postoperative nausea and vomiting Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Gastric volume | prior to anesthesia induction
  Assessment of gastric volume by ultrasound

SECONDARY OUTCOMES:
preoperative anxiety | before coming to the operating room, Scored between 20 and 80 points. A high score indicates high anxiety
  preoperative anxiety will be assessed with the State-Trait Anxiety Inventory
postoperative nausea and vomiting | up to postoperative 24 hours, numeric rank score is scored between 0 and 3 points
  postoperative nausea and vomiting scores of the patients will be evaluated
thirst, hunger, fatigue, dry mouth | before drink (2 hous before surgery), prior to anesthesia induction, visual analog scale is scored between 0 and 10
  thirst, hunger, fatigue, dry mouth will be evaluated with visual analog scale
Postoperative Pain Score | up to postoperative 24 hours, visual analog scale is scored between 0 and 10
  Postoperative Pain Score will be evaluated with visual analog scale
postoperative insulin resistance | glucose, insulin and cortisol will be measured 2 hours before surgery(before drink), before induction and 2 hours postoperatively
  Blood glucose mg/dL, Insulin milli-International unit/L, Cortisol µg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06289543/Prot_SAP_000.pdf